CLINICAL TRIAL: NCT07339670
Title: Effect of Smoking on the Expression of Periodontal Ligament -Associated Protien-1 and Sclerostin in Gingival Crevicular Fluid of Stage II Periodontitis Patients After Non-Surgical Periodontal t\Therapy
Brief Title: Study of Gum Tissue Proteins in Smokers vs. Non-smokers After Cleaning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Manar Morsi elsaied morsi, dentist, Al-Azhar University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OMPDR_105_1r
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Smoking ( Cigarette); Periodontitis Stage II
MeSH Terms: conditions — Cigarette Smoking; Periodontitis | interventions — Listerine; Ethanol; methyl salicylate; Menthol; Thymol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smoker with periodontitis (Active Comparator): patients with stage II periodontitis who are current smoker and will receive non-surgical periodontal therapy
  Interventions: Procedure: Non Surgical Periodontal Treatment includes post operative mouth wash with Listerine® (ethanol 21.6%, methyl salicylate 0.06%, menthol 0.042%, thymol 0.064% and eucalyptol 0.092%)
- Non-smokers with periodontitis (Active Comparator): patients with stage II periodontitis who have never smoked and will receive Non-surgical therapy
  Interventions: Procedure: Non Surgical Periodontal Treatment includes post operative mouth wash with Listerine® (ethanol 21.6%, methyl salicylate 0.06%, menthol 0.042%, thymol 0.064% and eucalyptol 0.092%)

INTERVENTIONS:
Procedure: Non Surgical Periodontal Treatment includes post operative mouth wash with Listerine® (ethanol 21.6%, methyl salicylate 0.06%, menthol 0.042%, thymol 0.064% and eucalyptol 0.092%) — scaling , curettage and root planning

SUMMARY:
The aim of this study is to evaluate how smoking affects the healing process of the gums after treatment. The researchers will measure the levels of two specific proteins (PLAP-1 and Sclerostin) in the gum fluid of patients with stage II periodontitis. These measurements will be compared between smokers and non-smokers before and after receiving non-surgical periodontal therapy (cleaning and scaling) to see if smoking changes the body's response to treatment.

DETAILED DESCRIPTION:
Patients diagnosed with Stage II Periodontitis will be recruited and divided into two groups: Group I (current smokers) and Group II (non-smokers). At the beginning of the study (baseline), clinical periodontal parameters will be recorded, including probing depth, clinical attachment level, and plaque index. Gingival Crevicular Fluid (GCF) samples will be collected from the most affected sites using paper strips.

Following the initial assessment, all participants will undergo non-surgical periodontal therapy consisting of full-mouth scaling and root planing (SRP) using ultrasonic and hand instruments. Oral hygiene instructions will be provided to all patients.

Patients will be re-evaluated after 6 months following the treatment. Clinical parameters will be re-recorded, and GCF samples will be collected again. The samples will then be analyzed using Enzyme-Linked Immunosorbent Assay (ELISA) to determine the concentration levels of Periodontal Ligament Associated Protein-1 (PLAP-1) and Sclerostin. The study aims to correlate these protein levels with the clinical healing outcomes in both smokers and non-smokers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged from 25 - 40 years old.
* Patients diagnosed as having Stage II periodontitis.
* Group of current smoker's patients, more than 10 cigarettes per day.
* Group of non-smoker's patients.
* Maximum probing depth ≤ 5 mm, mostly horizontal bone loss.
* Clinical Attachment loss from 3-4 mm.
* Radiographic bone loss about 15% to 33%, mostly horizontal.

Exclusion Criteria:

* Pregnant or lactating women.
* Any known systemic disease.
* Patients who received periodontal treatment in last 6 months.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
change in periodontal ligament associated protien-1 levels | Baseline (before treatment) and 6 months after treatment
  Concentration of PLAP-1 measured in Gingival Crevicular Fluid (GCF) using ELISA technique. This protein reflects the status of the periodontal ligament.
Change in Sclerostin levels | Baseline and 6 months after treatment
  Concentration of Sclerostin measured in Gingival Crevicular Fluid (GCF) to evaluate bone remodeling activity.

SECONDARY OUTCOMES:
Change in Probing Pocket Depth | Baseline , 3 and 6 months after treatment
  Measurement of the depth of the gum pockets using a periodontal probe to assess clinical healing.
Change in Clinical Attachment Level | Baseline , 3 and 6 months after treatment
  Measurement of the distance from the cemento-enamel junction to the bottom of the pocket to assess tissue attachment gain.
Change in Plaque Index (PI). | Baseline , 3 and 6 months after treatment.
  Evaluation of the amount of plaque on tooth surfaces using the Silness and Löe Plaque Index. Scores range from 0 (no plaque) to 3 (abundance of soft matter). Lower scores indicate better oral hygiene.
Change in Gingival Index (GI). | Baseline, 3 and 6 months after treatment.
  Assessment of the severity of gingival inflammation using the Löe and Silness Gingival Index. Scores range from 0 (normal gingiva) to 3 (severe inflammation, tendency to spontaneous bleeding).
Change in Bleeding on Probing (BOP) percentage. | Baseline, 3 and 6 months after treatment.
  Presence or absence of bleeding recorded within 30 seconds after probing. It is calculated as the percentage of sites that bleed upon probing relative to the total number of sites probed.

CONTACTS AND LOCATIONS:
Overall Officials: Manar Morsi Morsi, MSc, Study Director — Faculty of Dental Medicine for Girls, Al-Azhar University
Locations (1):
- Faculty of Dental Medicine for Girls, Al-Azhar University, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be available to preserve patient confidentiality and because the informed consent signed by participants did not include a provision for public data sharing